CLINICAL TRIAL: NCT05438784
Title: Comparison of Two Different Modalities for Orbital Reconstruction Based on CAD-CAM Technology: A Clinical Randomized Trial
Brief Title: Application of CAD-CAM Technology in Orbital Bone Reconstruction
Acronym: CAD-CAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hatem Adel Aboelhassan (Other)
Responsible Party: Sponsor-Investigator, Hatem Adel Aboelhassan, specialist of maxillofacial, head and neck surgery, Sohag University
Organization: Sohag University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-22-06-18
Record Dates: First submitted 2022-06-21; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Orbital Bone Fracture; Maxillary Cyst; Maxillary Neoplasms; Zygomatic Fractures; Orbital Neoplasms; Facial Deformity
Keywords: Orbital bone reconstruction; zygomaticomaxillary complex fracture (ZMC); patient specific implant; preformed plates; CAD-CAM
MeSH Terms: conditions — Orbital Fractures; Maxillary Neoplasms; Zygomatic Fractures; Orbital Neoplasms

STUDY DESIGN:
Intervention Model Description: the participants are assigned to two groups randomly A and B and receive two different intervention modality throughout the study and the results will be compared between the two groups
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (patient specific titanium implant) (Active Comparator): (reconstruction with patient specific titanium implant)
  Interventions: Procedure: orbital bone reconstruction with patient specific titanium implant
- Group B (preformed plate bended on stereolithographic model) (Active Comparator): (reconstruction with preformed titanium plate preoperatively bended on stereolithographic model)
  Interventions: Procedure: orbital bone reconstruction with preformed titanium plate preoperatively bended on stereolithographic model

INTERVENTIONS:
Procedure: orbital bone reconstruction with patient specific titanium implant — orbital defects reconstruction will be virtually planned by software and a patient specific titanium implant will be manufactured using milling technique depending on CAD-CAM technology
  Arms: Group A (patient specific titanium implant)
Procedure: orbital bone reconstruction with preformed titanium plate preoperatively bended on stereolithographic model — orbital defects reconstruction will be virtually planned by software and a reconstructed stereolithographic model will be 3D printed and used for preoperatively bending of preformed titanium implant.
  Arms: Group B (preformed plate bended on stereolithographic model)

SUMMARY:
Reconstruction of orbital defects resulting after trauma; tumor resection; maxillary cyst; craniofacial anomalies and sequestrated bone…. etc., has been a challenging issue over the years and this owing to the complicated anatomy of orbit. Inaccurate orbital reconstruction may lead to devastating cosmetic and functional complications. Titanium mesh for orbital reconstruction has now become "probably" the most popular material for orbital wall reconstruction worldwide. Innovation of CAD-CAM technology and its application in maxillofacial surgery will markedly improve the surgical outcome. This study will assess the accuracy of orbital reconstruction using CAD-CAM technology and to compare two different modalities for orbital reconstruction based on this technology.

DETAILED DESCRIPTION:
This study will be a prospective cohort study. It will include patients treated with the custom-made implants for orbital blow out fractures, ZMC fractures or tumors. The sample will consist of 34 patients who will need orbital reconstruction and will be operated in Maxillofacial, Head and Neck Unit, General Surgery Department, Faculty Of Medicine, Sohag University, Egypt. The patients will be randomly divided into two groups, group (A) reconstructed with patient specific implant and group (B) reconstructed with preformed plate preoperatively bended on stereolithographic model. The reconstructive outcomes are assessed by clinical and ophthalmological examinations and accuracy analysis by comparing the preoperative and postoperative multi slice computed tomography data. All patients will be assessed clinically, ophthalmologically, and radiographically using computed tomography (CT) then virtual surgical planning and custom-made patient implant will be manufactured. Post-operative clinical evaluation will be done, and radiographic evaluation of all patients will be done by CT scan within one week and 6 months after the procedure. comparing data of the two groups will be done using appropriate methods.

ELIGIBILITY:
Inclusion Criteria:

* fracture of the orbital floor and/or medial wall and/or lateral wall.
* complex fracture of the zygomatic bone (those affecting orbital volume).
* Old orbital fractures on either side causing enophthalmos, diplopia, cosmetic asymmetry.
* Periorbital neoplasm affecting orbital volume and need surgical resection

Exclusion Criteria:

* injury to the globe that restricts surgical reconstruction.
* neurological diseases with influence on eye motility or sight.
* Patients with special needs.
* Medically compromised patients who are not fit for surgery.
* Patients refused participation in this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
measurement of Changes in orbital bony volume | preoperative and one week and 6 months post-operative
  pre and post operative reconstructed orbit volume will be measured using multi slice computed tomography (MSCT) image loaded on software and compared with preoperative and with healthy non affected orbit

SECONDARY OUTCOMES:
measurement of Changes in globe position in the bony orbit | preoperative and one week and 6 months post operative
  pre and post operative measurement of globe position within the bony orbit using MSCT image loaded on software and comparing measures with preoperative and with healthy non affected orbit
measurement of Changes in zygomaticomaxillary complex symmetry | preoperative and one week and 6 months post operative
  in patients with associated ZMC affection, symmetry with the healthy side and prominence of the zygomatic eminence will be measured using MSCT image loaded on software and compared with preoperative and with healthy non affected ZMC

OTHER OUTCOMES:
changes in ocular motility pre and post-operative | preoperative and one week ,one month ,3rd and 6th month post operative
  assessment of motility of eye globe using extraocular muscle function test
cost of the implant in US dollar | Through study completion, an average of 1 year
  cost of the patient specific implant and the cost of the stereolithographic model and preformed titanium implant
adverse events | postoperative one week , 3rd and 6th moths postoperative
  implant displacement, bleeding, infection, pain
changes in patient satisfaction using scoring system from 1 to 5 | 1st, 3rd and 6th month post operative
  assessment of the patients satisfaction to the results post operative using scoring system from 1 to 5 in which :
  * 1 = Excellent
  * 2 = good
  * 3 = Fair
  * 4 = not bad
  * 5 = poor
duration of surgery | intraoperative
  recording each procedure time
measurement of changes in visual acuity using A Snellen chart test | preoperative and one week ,one month ,3rd and 6th month post operative
  testing of visual acuity of the affected eye pre and post operative
changes in aesthetic results using scoring system from 1 to 4 | 1st, 3rd and 6th month post operative
  assessment of changes in cosmetic results following surgery by one of the supervisors using a scoring system from 1 to 4 in which:
  * 1 = Excellent
  * 2 = good
  * 3 = Fair
  * 4 = poor

CONTACTS AND LOCATIONS:
Overall Officials: Kamal A Hassanein, Professor, Study Chair — Sohag University; Tarek A Ftohy, Ass. prof, Study Director — Sohag University; Islam AA Amer, Ass. prof, Study Director — Sohag University
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abbate V, Iaconetta G, Califano L, Pansini A, Bonavolonta P, Romano A, Salzano G, Somma T, D'Andrea L, Dell'Aversana Orabona G. Self-Made Rapid Prototyping Technique for Orbital Floor Reconstruction: Showcases for Technical Description. J Craniofac Surg. 2019 Oct;30(7):2106-2110. doi: 10.1097/SCS.0000000000006004. PMID 31513039
- [Background] Zimmerer RM, Ellis E 3rd, Aniceto GS, Schramm A, Wagner ME, Grant MP, Cornelius CP, Strong EB, Rana M, Chye LT, Calle AR, Wilde F, Perez D, Tavassol F, Bittermann G, Mahoney NR, Alamillos MR, Basic J, Dittmann J, Rasse M, Gellrich NC. A prospective multicenter study to compare the precision of posttraumatic internal orbital reconstruction with standard preformed and individualized orbital implants. J Craniomaxillofac Surg. 2016 Sep;44(9):1485-97. doi: 10.1016/j.jcms.2016.07.014. Epub 2016 Jul 21. PMID 27519662
- [Background] Felding UNA. Blowout fractures - clinic, imaging and applied anatomy of the orbit. Dan Med J. 2018 Mar;65(3):B5459. PMID 29510812
- [Background] Mustafa SF, Evans PL, Bocca A, Patton DW, Sugar AW, Baxter PW. Customized titanium reconstruction of post-traumatic orbital wall defects: a review of 22 cases. Int J Oral Maxillofac Surg. 2011 Dec;40(12):1357-62. doi: 10.1016/j.ijom.2011.04.020. Epub 2011 Aug 31. PMID 21885249
- [Background] Raisian S, Fallahi HR, Khiabani KS, Heidarizadeh M, Azdoo S. Customized Titanium Mesh Based on the 3D Printed Model vs. Manual Intraoperative Bending of Titanium Mesh for Reconstructing of Orbital Bone Fracture: A Randomized Clinical Trial. Rev Recent Clin Trials. 2017;12(3):154-158. doi: 10.2174/1574887112666170821165206. PMID 28828975
- [Background] Sugar AW, Kuriakose M, Walshaw ND. Titanium mesh in orbital wall reconstruction. Int J Oral Maxillofac Surg. 1992 Jun;21(3):140-4. doi: 10.1016/s0901-5027(05)80780-5. PMID 1640125
- [Background] Bly RA, Chang SH, Cudejkova M, Liu JJ, Moe KS. Computer-guided orbital reconstruction to improve outcomes. JAMA Facial Plast Surg. 2013 Mar 1;15(2):113-20. doi: 10.1001/jamafacial.2013.316. PMID 23306963
- [Background] Longeac M, Depeyre A, Pereira B, Barthelemy I, Pham Dang N. Virtual surgical planning and three-dimensional printing for the treatment of comminuted zygomaticomaxillary complex fracture. J Stomatol Oral Maxillofac Surg. 2021 Sep;122(4):386-390. doi: 10.1016/j.jormas.2020.05.009. Epub 2020 May 18. PMID 32439600
- [Background] Scolozzi P. Applications of 3D orbital computer-assisted surgery (CAS). J Stomatol Oral Maxillofac Surg. 2017 Sep;118(4):217-223. doi: 10.1016/j.jormas.2017.05.007. Epub 2017 Jun 19. PMID 28642192